CLINICAL TRIAL: NCT07004816
Title: The Mutation Profile and Prognosis in Acute Myeloid Leukemia With IDH1/2 Mutation
Brief Title: The Mutation Profile and Prognosis in AML With IDH1/2 Mutation
Status: Terminated | Type: Observational
Why Stopped: Adapted the plan
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2017004
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-05

CONDITIONS: AML

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML patients: Uncover mutation profiles of newly-diagnosed AML patients
  Interventions: Other: Uncover mutation profiles

INTERVENTIONS:
Other: Uncover mutation profiles — Uncover mutation profiles

SUMMARY:
Investigators have a prospective clinical cohort including 500 adult AML patients. And investigators have stored leukemia sample from these patients. In this program investigators will do mutation profile in these patients. Also, investigators will elucidate the incidence of IDH1/2 mutations in adult AML in China and elucidate the prognostic effect of IDH1/2 mutation in AML.

DETAILED DESCRIPTION:
In this program, first, investigators want to uncover mutation profiles in the 500 AML patients including AML1-ETO CBFb-MYH11, MLL translocation, NPM1, FLT3, DNMT3a, CEBPA, TET2, ASXL1, U2AF2, TP53, c-KIT, RUNX1, NRAS, KRAS, PTPN11 genetic alteration in addition to IDH1/2 mutation. These patients received regimen, which is consistent with NCCN and ELN guidelines. NPM1, FLT3, DNMT3a, CEBPA, TET2, ASXL1, U2AF2, TP53, c-KIT, RUNX1, NRAS, KRAS, PTPN11, and IDH1/2 genetic alteration will be detected by targeted next generation sequencing. AML1-ETO and CBFb-MYH11 will be detected by RT-PCR. MLL translocation will be detected by FISH(fluorescence in situ hybridization).Next, investigators will elucidate the incidence of IDH1/2 mutations in adult AML in China. Then investigators will investigate mutation profile in IDH1/2 mutation AML patients. Finally, investigators will elucidate the prognostic effect of IDH1/2 mutation in AML. At last, investigators will instigate how mutation profile affects the prognosis in IDH1/2 mutation AML patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age of less than 60 years old;
2. Patients that meet the diagnostic criteria(WHO 2008 criteria) of AML (except APL subtypes).
3. Adult patients are willing to participate in the study and sign the informed consent by themselves or by their immediate family. Patients under 18 years old willing to participate should have their legal guardians sign the informed consent.

Exclusion Criteria:

1. Patients with other blood diseases(for example, haemophiliacs) are excluded.
2. With mutation of breakpoint cluster region-Abelson(BCR-ABL) fusion gene and in need of tyrosine kinase inhibitors therapy;
3. Acute panmyelosis with myelofibrosis and myeloid sarcoma patients;
4. Had other malignant tumor in need of treatment;
5. Patients with other factors which were considered unsuitable to participate in the study by the investigators.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Investigators have a prospective clinical cohort including 500 adult AML patients. And investigators have stored leukemia sample from these patients. In this program investigators will do mutation profile in these patients. Also, investigators will elucidate the incidence of IDH1/2 mutations in adult AML in China and elucidate the prognostic effect of IDH1/2 mutation in AML.
Sampling Method: Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Incidence | Before treatment
  Incidence is defined as the incidence of patients who carries IDH1/2 mutations

SECONDARY OUTCOMES:
Relapse-Free Survival(RFS) | Up to 3 years
  RFS is defined as the time from the date of complete remission (CR) after entry in this trial until the date of documented relapse or death for subjects who achieve CR.
Overall Survival(OS) | Up to 3 years
  OS is defined as the time from the date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No